CLINICAL TRIAL: NCT05191043
Title: Effects of Kinesio Taping in Addition to Routine Physical Therapy on Pain, Range of Motion and Functional Disability in Patients With Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/998/2021
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Cervical Pain
Keywords: Upper Cross Syndrome; kinesio taping; Neck disability index; goniometer; pain
MeSH Terms: conditions — Neck Pain; Oculocerebral hypopigmentation syndrome type Preus; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A/ kinesio taping group (Experimental): Routine physical therapy along with Kinesio Taping
  Interventions: Other: Kinesio Taping Technique; Other: Routine Physical Therapy
- Group B/ routine physical therapy (Active Comparator): routine physical therapy
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Kinesio Taping Technique — Kinesio taping is a thin, stretchy, elastic cotton strip with an acrylic adhesive that is approximately the same thickness as the epidermis of the skin. When the taping method is followed correctly, the tape effects on the muscle by facilitating a weakened muscle or relaxing an over-used muscle,decreasing pain, fatigue and increasing tissue recovery. Kinesio Taping facilitation technique will be used with fifty percent stretch on rhomboids bilaterally.
  Arms: Group A/ kinesio taping group
Other: Routine Physical Therapy — routine physical therapy includes thermotherapy and Transcutaneous electrical nerve stimulation (TENS), the strengthening exercises of lower and middle trapezius, rhomboids and deep neck flexors. Stretching exercises of upper trapezius, pectoralis major and minor. Mobilization of cervicothoracic junction and postural education.
  Thermotherapy and transcutaneous electrical nerve stimulation will be used for 10 minutes in each session. Each exercise will be performed in 3 sets of 10 repetitions. Treatment session will have a duration of 30-45 minutes.

SUMMARY:
Objective of the study is to compare the effects of kinesio taping and routine physical therapy on pain, range of motion and functional disability in patients with upper cross syndrome.It is a single blinded randomized controlled trial using non probability purposive sampling technique.

ALTERNATIVE HYPOTHESIS:

There is a significant difference in the effects of routine physical therapy with and without kinesio taping on pain, range of motion and functional disability in patients with upper cross syndrome.

NULL HYPOTHESIS:

There is no significant difference in the effects of routine physical therapy with and without kinesio taping on pain, range of motion and functional disability in patients with upper cross syndrome.

DETAILED DESCRIPTION:
It will be a prospectively registered ,parallel designed, randomized controlled trial with concealed allocation. Subjects will be selected from the outpatient Department of Physical Therapy, The University of Lahore Teaching Hospital,Lahore, Pakistan. Patients who met eligibility criteria will be informed about the aim of study.all the eligible participants who will agree to participate will sign a consent form. After baseline assessment selected participants will be divided into 2 groups by random allocation method.Subjects will be randomized into two groups using computer generated random numbers.The outcome assessor will be unaware of treatment given to both groups.The calculated sample size using Numeric pain rating scale as outcome measure is 28 in each group, but after adding 20% dropout, the sample size will be 28+6=34 in each group, allowing statistical power of 80%and alpha level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Participants with an age between 18 to 40
* Participants diagnosed with chronic upper cross syndrome by orthopedic department for physical therapy treatment

Exclusion Criteria:

* Trauma, Tumor and Fracture of upper limb and shoulder
* Congenital deformities of upper limb
* History of any systemic disease
* History of any neurological disease (epilepsy &seizure, Parkinson's disease)
* History of recent surgery of spine or shoulder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale( assessing change in pain at between baseline, at 1st week, 2nd week and at the end of 4th week of treatment) | baseline, 1st week ,2nd week and 4th week
  This is 11 points scale ranges from 0-10, where 0 means no pain and 10 is the worst pain. The values ranges from 1-3 means mild pain; 4-6 is considered moderate pain; 7-10 is severe pain. the average of three readings is considered as pain value.
Universal Goniometer (to assess change in range of motion at baseline,1st,2nd and 4th week.) | baseline, 1st week ,2nd week and 4th week
  A universal goniometer is a device that measures an angle or permits rotation of an object to a definite position. It is designed like a protractor and may form a full or a half-circle from 0 to 180 degrees or 180 to 0 degrees for half circle models or 0 to 360 degrees on full circle.Normal range of motion of flexion 0-45 ₒ extension, 0-45 ₒ, side flexion 0-45 ₒ , rotation 0-80.
Neck disability Index ( assessing change in neck functional activities at baseline, 1st,2nd and 4th week) | baseline, 1st,2nd and 4th week
  This is the Patient-completed, condition-specific functional status questionnaire with 10 items for measuring disability in patients with neck pain.It contains 10 pain-related questions scored from 0 (no pain) to 5 (most severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Ghafoor, MSPT, Principal Investigator — University of Lahore
Locations (1):
- Waqar Afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No